CLINICAL TRIAL: NCT00004012
Title: A Phase II Trial of Oral Capecitabine in Patients With Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma
Brief Title: Capecitabine in Treating Patients With Recurrent Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-112; CDR0000067229 (Registry Identifier: PDQ (Physician Data Query)); NCI-G99-1556
Record Dates: First submitted 1999-11-01; First posted 2004-05-25 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Capecitabine

INTERVENTIONS:
Drug: capecitabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of capecitabine in treating patients who have recurrent ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and time to treatment failure in patients with recurrent ovarian epithelial, fallopian tube, or primary peritoneal carcinoma treated with oral capecitabine. II. Determine the tolerability and safety of this regimen in these patients.

OUTLINE: Patients receive oral capecitabine twice daily for 14 days. Treatment continues every 3 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 14-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent ovarian epithelial carcinoma, fallopian tube cancer, or primary peritoneal cancer previously treated with at least one cisplatin based chemotherapy regimen Prior repeat treatment with a taxane and/or platinum agent allowed Prior repeat treatment with other chemotherapy agent allowed once Recurrent disease defined as: At least one site of measurable disease by radiograph and/or a rise of CA-125 over a minimum of 3 samples to a level of at least 50% of upper limit of normal

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 2.0 times upper limit of normal (ULN) SGOT less than 2.0 times ULN Alkaline phosphatase less than 2.0 times ULN Renal: Creatinine no greater than 1.5 mg/dL Other: Must be able to take oral medication

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No prior fluorouracil based chemotherapy Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-12; Primary Completion 2000-12 (Actual); Study Completion 2000-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sabbatini, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States